CLINICAL TRIAL: NCT03933956
Title: Metabolic Effects of the SGLT-2 Inhibitor Empagliflozin in Patients With Diabetic Nephropathy (MEDiaN)
Acronym: (MEDiaN)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated owing to challenges posed by the COVID-19 situation.
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEDiaN2018; Duke-NUS-TIDR/2018/0010 (Other Grant/Funding Number: Tanoto Initiative for Diabetes Research Award)
Record Dates: First submitted 2019-04-20; First posted 2019-05-01 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetic nephropathy; Sodium-glucose Cotransporter 2 Inhibitors
MeSH Terms: conditions — Diabetic Nephropathies | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single-arm open-label intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin-treated (Experimental): Oral empagliflozin tablets 10mg daily, taken for 30 days.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Oral empagliflozin 10mg daily for 30 days
  Other Names: Jardiance

SUMMARY:
The MEDiaN study aims to examine the state of fuel metabolism in participants with diabetic nephropathy (DN) before and after the use of the sodium-glucose transport protein 2 inhibitor (SGLT-2i) empagliflozin. The goals of the MEDiaN study are to better understand the contribution of fuel metabolism to the development of DN, and to determine if changes to fuel metabolism can have a positive impact on this disease.

The MEDiaN study is a single-center single-arm open-label intervention study to examine the effects of empagliflozin 10mg daily taken for 30 days on fuel oxidation patterns in participants with type 2 diabetes and DN.

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is a common cause of end-stage renal disease. MEDiaN study investigators hypothesize that dysregulated mitochondrial fuel oxidation is a major driver of diabetic nephropathy. The sodium-glucose transport protein 2 inhibitor (SGLT-2i) empagliflozin has been shown to slow the progression of DN in patients with diabetes.

The MEDiaN study aims to examine the state of fuel metabolism in participants with DN before and after the use of the SGLT-2i empagliflozin. The goals of the MEDiaN study are to better understand the contribution of fuel metabolism to the development of DN, and to determine if changes to fuel metabolism can have a positive impact on this disease.

The MEDiaN study is a single-center single-arm open-label intervention study to examine the effects of empagliflozin 10mg daily taken for 30 days on fuel oxidation patterns in participants with type 2 diabetes and DN.

The MEDiaN study plans to recruit 40 participants aged 21 to 100 years of age with type 2 diabetes mellitus and diabetic nephropathy. Participants will receive treatment with oral empagliflozin 10mg daily for 30 days. The state of fuel metabolism will be examined through metabolomics analysis of blood and urine samples before and after empagliflozin 10mg daily taken for 30 days.

ELIGIBILITY:
Inclusion criteria:

1. Man or woman between 21 and 100 years of age
2. Type 2 diabetes mellitus as defined by:

   * Fasting plasma glucose ≥7.0mmol/l, or
   * Symptoms of hyperglycemia with casual plasma glucose ≥11.1 mmol/L, or
   * 2-hour plasma glucose ≥11.1 mmol/l after a 75-gram oral glucose load, or
   * Known type 2 diabetes mellitus diagnosed by a medical practitioner
3. Two or more measurements indicating increased urine protein excretion within 1-year

   Increased urine protein excretion is defined as:
   * Urine microalbumin/creatinine ratio (ACR) > 3.3 mg/mmol creatinine or
   * Urine total protein/creatinine ratio (PCR) > 0.2 g/urine creatinine
4. Known diabetes duration > 3 months
5. HbA1c ≤9% (within 3 months prior to enrolment)
6. Not currently treated with an SGLT-2 inhibitor, and have not received SGLT-2 inhibitor therapy within the last 10 weeks.
7. Stable diabetes therapy for at least 3months as defined as:

   * No increase in dose of diabetes medications by more than two-fold or
   * No new agents added within the previous 3 months
8. Stable doses of angiotensin converting enzyme (ACE) inhibitors or angiotensin AT(1)-receptor blockers (ARBs) for at least 3 months.
9. Capable of providing informed consent

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Ketosis-prone diabetes
3. Previous diabetic ketoacidosis
4. History of Fournier's gangrene or skin and soft tissue infections of the perineum
5. Recurrent or severe urinary tract or genital mycotic infections, or history of genitourinary infection within 2 weeks prior to informed consent
6. Significant renal impairment (estimated Glomerular Filtration Rate < 45 ml/min/1.73m2**)
7. Dialysis or kidney transplant
8. Renal artery stenosis
9. Alanine aminotransferase or aspartate aminotransferase above 3x upper limit of normal
10. Significant change in weight (≥10% in the preceding 6 months)
11. Treatment with anti-obesity drugs
12. Previous bariatric surgery or other gastrointestinal surgeries that induce chronic malabsorption
13. Treatment with systemic glucocorticoids
14. Blood dyscrasias or clinically significant anaemia (Haemoglobin < 10 g/L)
15. Medical condition likely to limit survival to less than 3 years
16. Uncontrolled thyrotoxicosis, untreated hypothyroidism
17. Any ongoing acute medical illnesses
18. Hospitalization within 1 month prior to enrolment
19. Nursing mothers
20. Pregnancy, currently trying to become pregnant, or of child-bearing potential and not practicing an acceptable method of birth control or do not plan to continue using this method throughout the study
21. Excessive alcohol intake (> 1 unit per day for women and > 2 units per day for men)
22. History of drug abuse
23. Pancreatic insulin deficiency from any cause (history of pancreatitis, pancreatic surgery)
24. Known intolerance or allergic reactions to empagliflozin or other SGLT-2 inhibitors
25. Current participation in another clinical trial, or ingestion of investigational drug in another trial within 30 days prior to enrolment.
26. Presence of any non-DN renal glomerular disease (e.g. IgA nephropathy, lupus nephritis, membranous glomerulonephritis, focal segmental glomerular sclerosis)
27. Any previous organ transplantation
28. Any factors likely to limit adherence to interventions (e.g. dementia; alcohol or substance abuse; history of unreliability in medication taking or appointment keeping; significant concerns about participation in the study from spouse, significant other or family members)
29. Failure to obtain informed consent from participant
30. Presence of postural hypotension or clinically significant dehydration (reduced skin turgor, dry oral mucosa, hypotension)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in lipid metabolome signature | Baseline and after 30 days of treatment with empagliflozin 10mg daily
  Change in lipid metabolome signature following 30 days of empagliflozin treatment
Change in ketone signature | Baseline and after 30 days of treatment with empagliflozin 10mg daily
  Change in ketone signature following 30 days of empagliflozin treatment
Change in amino acid metabolome signature | Baseline and after 30 days of treatment with empagliflozin 10mg daily
  Change in amino acid metabolome signature following 30 days of empagliflozin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yun Rui Amanda Lam, MBBS MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu JJ, Ghosh S, Kovalik JP, Ching J, Choi HW, Tavintharan S, Ong CN, Sum CF, Summers SA, Tai ES, Lim SC. Profiling of Plasma Metabolites Suggests Altered Mitochondrial Fuel Usage and Remodeling of Sphingolipid Metabolism in Individuals With Type 2 Diabetes and Kidney Disease. Kidney Int Rep. 2016 Dec 16;2(3):470-480. doi: 10.1016/j.ekir.2016.12.003. eCollection 2017 May. PMID 29142974
- [Background] Sharma K, Karl B, Mathew AV, Gangoiti JA, Wassel CL, Saito R, Pu M, Sharma S, You YH, Wang L, Diamond-Stanic M, Lindenmeyer MT, Forsblom C, Wu W, Ix JH, Ideker T, Kopp JB, Nigam SK, Cohen CD, Groop PH, Barshop BA, Natarajan L, Nyhan WL, Naviaux RK. Metabolomics reveals signature of mitochondrial dysfunction in diabetic kidney disease. J Am Soc Nephrol. 2013 Nov;24(11):1901-12. doi: 10.1681/ASN.2013020126. Epub 2013 Oct 10. PMID 23949796
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Perrone-Filardi P, Avogaro A, Bonora E, Colivicchi F, Fioretto P, Maggioni AP, Sesti G, Ferrannini E. Mechanisms linking empagliflozin to cardiovascular and renal protection. Int J Cardiol. 2017 Aug 15;241:450-456. doi: 10.1016/j.ijcard.2017.03.089. Epub 2017 Mar 23. PMID 28395981
- [Background] Mudaliar S, Alloju S, Henry RR. Can a Shift in Fuel Energetics Explain the Beneficial Cardiorenal Outcomes in the EMPA-REG OUTCOME Study? A Unifying Hypothesis. Diabetes Care. 2016 Jul;39(7):1115-22. doi: 10.2337/dc16-0542. PMID 27289124
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454

DOCUMENTS (1):
  • Study Protocol (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03933956/Prot_000.pdf